CLINICAL TRIAL: NCT01616550
Title: Quality of Postoperative Pain Management Following Thoracic Surgery: a Prospective Observational Study.
Brief Title: Quality of Postoperative Pain Management Following Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: DB 2012-001
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Postoperative Pain
Keywords: analgesia; thoracic surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesia; Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing thoracic surgery: Assessment of postoperative pain management in patients undergoing elective thoracoscopy or thoracotomy in a teaching hospital
  Interventions: Other: Assessment of pain using the Brief Pain Questionnaire; Other: Assessment of pain relief using a Verbal Numeric Scale (VNS); Other: Assessment of patient' satisfaction with pain relief; Other: Nurse's satisfaction with patient's pain relief and recovery

INTERVENTIONS:
Other: Assessment of pain using the Brief Pain Questionnaire — Patients will complete this questionnaire daily from surgery until discharge from the hospital
Other: Assessment of pain relief using a Verbal Numeric Scale (VNS) — Patients will assess their pain daily from surgery until discharge from the hospital using the VNS
Other: Assessment of patient' satisfaction with pain relief — Will be assessed three times a day using a scale from 1 to 4 (1= very unsatisfied, 4= very satisfied)
Other: Nurse's satisfaction with patient's pain relief and recovery — Will be assessed three times a day using a scale from 1 to 4 (1= very unsatisfied, 4= very satisfied)

SUMMARY:
The purpose of this study is to assess the quality of postoperative pain management in a Canadian teaching hospital following thoracic surgery.

Hypothesis: Postoperative pain management following thoracotomy or thoracoscopy is still suboptimal despite the evidence that adequate pain relief improves outcome.

DETAILED DESCRIPTION:
Pain is an expected outcome of surgery. However, many patients experience suboptimally managed postoperative pain. Benefits of adequate analgesia no longer need to be demonstrated. Optimal analgesia leads to faster recovery, reduces the risk of postoperative complications, enhances patient's satisfaction and quality of life following surgery.

Currently, approximately 1000 thoracic surgeries are performed in our hospital annually. Many of these surgeries that previously required a thoracotomy incision are now performed under Video-Assisted Thoracoscopy Surgery (VATS). Although VATS is known to be less invasive and causes less pain than thoracotomy, some patients still experience considerable pain following thoracoscopy especially during the first hours following surgery.

Thoracic epidural has emerged as the preferred pain control technique following thoracotomy. However, the role of epidural analgesia after thoracoscopy remains debatable. The ideal postoperative analgesia regimen for the short-duration but intense pain related to thoracoscopy has not been elucidated. Paravertebral blockade is an alternative to epidural analgesia. However, the duration of pain relief associated with this technique may vary from 4 to 48 hours. Systemic opioids given through patient-controlled devices may be used after thoracic surgery but the analgesic effect can be limited and undesirable side-effects may occur.

This prospective observational study will investigate the quality of pain management following thoracic surgery and assess patient's and nurse's satisfaction regarding pain relief in a teaching hospital.

Methods:

Patients scheduled for elective thoracic surgery to be performed by thoracotomy or thoracoscopy will be considered for this prospective observational study.

The surgical approach and pain management plan will not be modified by the patient's participation to the study. According to standard practice in our hospital, pain will be assessed using a Verbal Numeric Scale from 0 to 10.

Type of analgesic technique, consumption of opioid and non-opioid drugs, type and duration of surgery will be noted. Side-effects attributable to analgesia and associated treatment will be recorded. Length of stay in the recovery room, step-down unit and in the hospital will also be recorded. Postoperative complications will be assessed.

Patients will be invited to complete the short form of the "Brief Pain Inventory". They will be asked to grade their satisfaction with pain relief using a scale from 1 to 4 (1= very unsatisfied, 4= very satisfied). Nurses will be asked to provide their opinion on patient's pain relief, ability to move and collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients aged 18-80 years
* ASA physical status 1-3
* Patients undergoing elective thoracic surgery (thoracotomy/thoracoscopy)

Exclusion Criteria:

* Current regular use of drugs belonging to the class of opioids
* Presence of a coexisting chronic pain syndrome
* The inability to understand a verbal numeric pain scale (VNS) despite previous instruction
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective thoracotomy or thoracoscopy in a teaching hospital over a one year period will be considered for this study
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain relief according to analgesic technique | From surgery (Day 0) until discharge from the hospital (Day 5)

SECONDARY OUTCOMES:
Consumption of analgesics | From surgery (Day 0) until discharge from the hospital (Day 5)
Interference of pain on daily activities | From surgery (Day 0) until discharge from the hospital (Day 5)
Patient's satisfaction with pain relief | From surgery (Day 0) until discharge from the hospital (Day 5)
Nurse's satisfaction with patient's pain relief, mobility and collaboration | From surgery (Day 0) until discharge from the hospital (Day 5)
Length of stay in the recovery room | From arrival (Day 0) until discharge from the recovery room (Day 0)
Length of stay in the step-down unit | From arrival (Day 0) until discharge from the step-down unit (Day 1)
Length of stay in the hospital | From surgery (Day 0) until discharge from the hospital (Day 5)
Side-effects attributable to analgesia | From surgery (Day 0) to discharge from the hospital (Day 5)
Presence of postoperative complications | From surgery (Day 0) until discharge from the hospital (Day 5)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Boudreault, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada